CLINICAL TRIAL: NCT02005250
Title: Bone Structure and Strength Evaluated by Extreme-CT Scan Before and After Treatment of Hyper- and Hypothyroidism
Status: Completed | Type: Observational
Sponsor: Steen Bonnema (Other)
Responsible Party: Sponsor-Investigator, Steen Bonnema, Consultant, phd, DMsc, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: Thyroid Xtreme
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Hyperthyroidism; Hypothyroidism
Keywords: osteoporosis; hyperthyroidism; hypothyroidism
MeSH Terms: conditions — Hyperthyroidism; Hypothyroidism; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hyperthyroidism: 61 pre- and postmenopausal women with hyperthyroidism
- hypothyroidism: 32 pre- and postmenopausal women with hypothyroidism

SUMMARY:
The aim to evaluate the bone structure by Dexa-scan, extreme CT and bone markers before and one year after treatment for a thyroid functional disorder

DETAILED DESCRIPTION:
The aim to evaluate the bone structure by Dexa-scan, extreme CT and bone markers before and one year after treatment for a thyroid functional disorder. Women with hyper- og hypothyroidism are included and undergo usual treatment. Patients are stratified into 10 different groups.

ELIGIBILITY:
Inclusion Criteria:

informed consent, female sex, age 20-85 years, indication for treatment of the thyroid disorder,

Exclusion Criteria:

pregnancy, renal insufficiency, known osteoporosis, other disease that may affect bone metabolism, medication which affects bone metabolism, T-score below -3.5, thyroidea ophthalmopathy with indication for steroids,

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with untreated hyper- or hypothyroidism
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2012-02; Primary Completion 2016-10 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steen Bonnema, phd, DMsci, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vinther CJ, Poulsen LH, Nicolaisen P, Obling ML, Brix TH, Hermann AP, Hegedus L, Jorgensen NR, Hansen S, Bonnema SJ. Do bone turnover markers reflect changes in bone microarchitecture during treatment of patients with thyroid dysfunction? J Endocrinol Invest. 2023 Feb;46(2):345-358. doi: 10.1007/s40618-022-01907-2. Epub 2022 Sep 5. PMID 36064878
- [Derived] Larsen CB, Riis KR, Winther KH, Larsen EL, Ellervik C, Hegedus L, Brix TH, Poulsen HE, Bonnema SJ. Treatment of Hyperthyroidism Reduces Systemic Oxidative Stress, as Measured by Markers of RNA and DNA Damage. J Clin Endocrinol Metab. 2021 Jun 16;106(7):e2512-e2520. doi: 10.1210/clinem/dgab273. PMID 33901280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients are enrolled consecutively, until maximum 200 participants are reached, or further enrollment is terminated on the decision by the sponsor.
Groups:
- Hyperthyroidism: 46 women with Graves' disease, toxic nodular goiter or subclinical hyperthyroidism
- Hypothyroidism: 27 women with overt or subclinical autoimmune hypothyroidism
Period: Overall Study
Arm/Group | Hyperthyroidism | Hypothyroidism
Started | 61 | 32
Completed | 46 | 27
Not Completed | 15 | 5
Not completed — Lost to Follow-up | 15 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperthyroidism | Hypothyroidism | Total
Number analyzed (Participants) | 46 | 27 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.83 (11.47) | 48.3 (11.3) | 53 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 27 | 73
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 46 | 27 | 73
Cortical thickness [Median (Inter-Quartile Range); unit: mm] | 0.74 [0.61 to 0.83] | 1.15 [1.01 to 1.24] | 0.90 [0.61 to 1.24]

OUTCOME MEASURES:

1. Primary Outcome: Thyroid Extreme CT
Description: Bone cortical thickness in the radius measured by high-resolution peripheral quantitative CT, in newly diagnosed thyroid disorder, before and after treatment aimed to obtain euthyroidism
Time Frame: one year
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Hyperthyroidism | Hypothyroidism
Number analyzed (Participants) | 46 | 27
mm | 0.89 [0.80 to 1.04] | 1.16 [1.02 to 1.32]

ADVERSE EVENTS:
Time Frame: 19 month
Description: Prospective monitoring and data collection of out-hospital patients during the study period
Arm/Group | Hyperthyroidism | Hypothyroidism
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/27
Other Adverse Events (participants affected / at risk) | 0/46 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No